CLINICAL TRIAL: NCT03358043
Title: Prevalence and Outcome of Acute Hypoxemic Respiratory Failure in Wales
Acronym: PANDORAWALES
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Jesus Villar, Clinical Scientist, Dr. Negrin University Hospital
Other Study IDs: ACPVM170916
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Acute Respiratory Insufficiency
Keywords: respiratory failure; mechanical ventilation; prevalence
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration, Artificial; Interactive Ventilatory Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mechanical ventilation — Consecutive intubated pateints receiving mechanical ventilation with a PaO2/FiO2≤300 mmHg on positive end-expiratory pressure (PEEP) of 5 cmH2O or more and FiO2 of 0.3 or more.
  Other Names: ventilatory support

SUMMARY:
This study is aimed to establish the epidemiological chacacteristics and clinical outcomes of mechanically ventilated patients with acute hypoxemic respiratory failure admitted in a network of hospitals from Wales (U.K.).

DETAILED DESCRIPTION:
The present study is aimed to establish the epidemiological characteristics and clinical outcomes of adult mechanically ventilated patients with acute hypoxemic respiratory failure [defined as a PaO2/FiO2 ≤300 mmHg on positive end-expiratory pressure (PEEP) of 5 cmH2O or more and FiO2 of 0.3 or more] admitted in a network of hospitals from Wales (U.K.). Although there are few previous published observational studies examining the incidence and mortality of patients with acute respiratory failure and ARDS, there are no studies specifically assessing the epidemiological characteristics, patterns of ventilation and clinical outcomes in patients with acute hypoxemic respiratory failure in the current era of lung protective ventilation. This study will be done simultaneously with the PANDORA (NCT03145974) in Spain.

The study is aimed to improve the knowledge on the epidemiology and outcome of ventilated patients, to identify the percentage of patients developing ARDS under the current definition, to validate a bedside scoring system for stratification of lung severity, and to examine the prognosis of hypoxemic respiratory failure, and risk factors associated with fatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18-year old.
* Endotracheal intubation and mechanical ventilation, independent of whether the need for ventilatory support is shorter or longer than 24 hours. Only patients receiving invasive mechanical ventilation can be included, although patients could have been on non-invasive ventilation before intubation.
* PaO2/FiO2 ≤300 mmHg on invasive mechanical ventilation with a PEEP of 5 cmH2O or more, and with a FiO2 of 0.3 or more.

Exclusion Criteria:

* No patients shhould be excluded (if they meet all the inclusion criteria), regardless of the underlying disease, estimated life expectancy, or duration of invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to participating ICUs will be screened daily. Only patients meeting inclusion criteria for acute hypoxemic respiratory failure will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypoxemic acute respiratory failure | 4 months
  The investigators will calculate the prevalence in relation to: (i) total number of ICU admissions; (ii) total number of mechanically ventilated patients during the study period; and (iii) per ICU bed available over the study period.

SECONDARY OUTCOMES:
Death in the hospital | Hospital stay (maximum 6 months)
  outcome before discharge to home (overall and in each category of acute hypoxemic respiratory failure)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, Study Chair — Clinical Scientist; Robert M Kacmarek, PhD, Study Chair — Clinical Scientist
Locations (12):
- United Kingdom (12):
  - Nevill Hall Hospital, Abergavenny
  - Ysbyty Gwynedd, Bangor
  - Cardiff University, Cardiff
  - University Hospital of Wales, Cardiff
  - Glangwili General Hospital, Carmarthen
  - Withybush General Hospital, Haverfordwest
  - Royal Glamorgan Hospital, Llantrisant
  - Prince Charles Hospital, Merthyr Tydfil
  - Royal Gwent Hospital, Newport
  - Ysbyty Glan Clwyd, Rhyl
  - Morriston Hospital, Swansea
  - Wrexham Maelor Hospital, Wrexham

IPD SHARING:
Plan to Share IPD: Undecided
Data from all patients must be collected and pooled by the coordinating center (Dr. Tamas Szakmany, All Wales Critical Care and Trauma Network)